CLINICAL TRIAL: NCT05436626
Title: Post-cholecystectomy Major Bile Duct Injury: Ideal Time to Repair Based on a Multicenter Study With Promising Results.
Brief Title: Post-cholecystectomy Major Bile Duct Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed Ahmed Omar, MD, Associate professor of surgery, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SVU/MED/SUR011/4/22/11/489
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Common Bile Duct Injury
Keywords: bile duct injury; reconstruction time; abdominal sepsis
MeSH Terms: conditions — Intraabdominal Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Early BDI reconstruction without abdominal sepsis control (Experimental): BDI reconstruction within 6 weeks after the injury without controlling the abdominal sepsis
  Interventions: Procedure: Early BDI reconstruction without abdominal sepsis control
- Early BDI reconstruction with abdominal sepsis control (Experimental): BDI reconstruction within 6 weeks after the injury after controlling the abdominal sepsis
  Interventions: Procedure: Early BDI reconstruction with abdominal sepsis control
- Delayed reconstruction (Active Comparator): BDI reconstruction after 6 weeks after the injury a
  Interventions: Procedure: Delayed reconstruction

INTERVENTIONS:
Procedure: Early BDI reconstruction without abdominal sepsis control — BDI reconstruction within 6 weeks after the injury without abdominal sepsis control
  Arms: Early BDI reconstruction without abdominal sepsis control
Procedure: Early BDI reconstruction with abdominal sepsis control — BDI reconstruction within 6 weeks after the injury with abdominal sepsis control
  Arms: Early BDI reconstruction with abdominal sepsis control
Procedure: Delayed reconstruction — BDI reconstruction after 6 weeks after the injury
  Arms: Delayed reconstruction

SUMMARY:
Bile duct injury (BDI) is one of the devastating recognized complications of cholecystectomy which does not respect the seniority or experience of the surgeon. It has a disastrous impact on long-term survival, health-related quality of life, and healthcare costs as well as high rates of litigation. The incidence of BDI increased with the introduction of laparoscopic cholecystectomy (LC) with an incidence of around 0.3-1.5%.

The initial aim of BDI is to manage abdominal and biliary sepsis and to transform an acute BDI into a controlled external biliary fistula.

The surgical treatment of postcholecystectomy BDI success depends on many factors as the severity of the injury, the centers and surgeon's experiences, the patient's condition, and the reconstruction time. The optimal time for the reconstruction and the patient's condition remains an active topic of interest and debate. Many papers discussed their impact on the short and long-term outcomes with different conflicting results from different institutions.

Based on the previous data and the absence of guidelines that recommend the timing of BDI reconstruction, the decision for the timing of reconstruction should be based on the predicted success of the operation, costs, and patient quality of life. If comparable morbidity and mortality outcomes can be obtained, patient quality of life and effective use of healthcare resources should be taken into consideration. We hypothesized that inadequate sepsis control and BDI reconstruction can be done safely at any time of presentation.

Our study aimed to present our experience in the management of major post-cholecystectomy BDI with HJ and analyze the impact of both the reconstruction time and the control of sepsis on the BDI reconstruction success rate. By analyzing the results of these three treatment strategies, we can better understand the factors that affect reconstruction success, costs, and health-related quality of life associated with BDI and subsequent repair.

DETAILED DESCRIPTION:
Bile duct injury (BDI) is one of the devastating recognized complications of cholecystectomy which does not respect the seniority or experience of the surgeon. It has a disastrous impact on long-term survival, health-related quality of life, and healthcare costs as well as high rates of litigation. Most of these patients are young females, between the ages of 30 and 50 years, with a long life expectancy, and in their most productive years. The incidence of BDI increased with the introduction of laparoscopic cholecystectomy (LC) with an incidence of around 0.3-1.5%; additionally, it results in complete transection. In Egypt, LC is developing rapidly in the primary hospitals that have bad medical conditions and the practicing surgeons have now still beyond the initial learning curve associated with this technique. As a result, the incidence of BDI increased, furthermore the majority were major and complex injuries. Based on the worldwide cholecystectomy frequency, even this low rate of BDI presents a significant potential healthcare burden. Due to this, it is critical that these patients have prompt recognition of their problem and reliable treatment with a long-term success rate. The initial aim of BDI is to manage abdominal and biliary sepsis and to transform an acute BDI into a controlled external biliary fistula. Following this, the severity of the damage should be evaluated. Whereas minor injuries are usually treated with endoscopic or percutaneous intervention, major injuries represent a major challenge even for hepatobiliary surgeons (HBS), and reconstructive surgery by hepaticojejunostomy (HJ) is usually indicated. Successful surgical reconstruction of Type E injuries can be as high as 90% when performed in highly specialized centers with expert multidisciplinary teams. Unfortunately, a considerable number of BDIs are still managed by injuring non-specialized surgeons in non-tertiary centers with poor surgical outcomes.

The surgical treatment of postcholecystectomy BDI success depends on many factors as the severity of the injury, the centers and surgeon's experiences, the patient's condition, and the reconstruction time. The optimal time for the reconstruction and the patient's condition remains an active topic of interest and debate. Many papers discussed their impact on the short and long-term outcomes with different conflicting results from different institutions.

Theoretically, intra-operative reconstruction of fresh injuries allows an adequate anastomosis and will be associated with the best surgical outcomes. But this is only feasible when BDI is recognized intraoperatively with a surgeon who has sufficient experience to carry out this repair. In most cases, this is far from being the case and is difficult to achieve either due to a small portion of BDIs that is diagnosed intraoperatively or the injuring surgeon who lacks sufficient experience to execute the repair that is almost always going to make an already challenging clinical situation worse.

For postoperative recognized BDI and contrary to the desire of most surgeons, most patients prefer early surgical repair. Early reconstruction (before 6 weeks) may have benefits in terms of reduced burden for the patient and the primary surgeon, avoiding re-admissions, improving patients' quality of life, and decreasing the total healthcare cost. Nevertheless, early reconstruction by which time the patient may be associated with severe local and systemic sepsis, hypoalbuminemia, and friable edematous non-dilated common bile duct (CBD) stump is not preferred by many surgeons for fear of anastomotic failure and bad surgical outcomes. In addition, at the time of an early repair, bile duct ischemia might still be developing, which could later result in anastomotic stricture, especially with associated vascular injuries. On the other hand, many surgeons prefer delayed repair (after 6 weeks) in a less inflamed surgical site with a more defined and properly vascularized duct stump without active sepsis. Taking into consideration that delayed reconstruction may require frequent procedures and repeated admissions as preoperative optimization with subsequent longer total in-hospital stay and increased total healthcare cost. In addition to the difficulty to convince most patients to wait for the delayed reconstruction and its benefits. Recently, many recent papers reported a significant association between adequate preoperative control of abdominal sepsis and reconstruction success rate with no impact of the BDI reconstruction time on the success rate.

Based on the previous data and the absence of guidelines that recommend the timing of BDI reconstruction, the decision for the timing of reconstruction should be based on the predicted success of the operation, costs, and patient quality of life.

If comparable morbidity and mortality outcomes can be obtained, patient quality of life and effective use of healthcare resources should be taken into consideration. We hypothesized that inadequate sepsis control and BDI reconstruction can be done safely at any time of presentation.

Our study aimed to present our experience in the management of major post-cholecystectomy BDI with HJ and analyze the impact of both the reconstruction time and the control of sepsis on the BDI reconstruction success rate. By analyzing the results of these three treatment strategies, we can better understand the factors that affect reconstruction success, costs, and health-related quality of life associated with BDI and subsequent repair.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with BDI within 6 weeks after open or laparoscopic cholecystectomy,
2. E1 to E4 BDI,
3. Failed stenting with endoscopic retrograde cholangiopancreatography (ERCP),
4. American Society of Anesthesiologists (ASA) score I-III,
5. Agreement to complete the study

Exclusion Criteria:

1. Advanced liver cirrhosis.
2. Benign or malignant bile duct stricture.
3. concomitant vascular and visceral injury

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Reconstruction success rate | 3 month
  The successful reconstruction was defined as the repair with HJ with no further intervention

SECONDARY OUTCOMES:
Operative time | 5 hours
  The time from skin incision to closure
Blood loss | 5 hours
  the total amount of blood loss during the operation
External stent | 90 days
  The use of external stent for the hepaticojejunostomy reconstruction
Drain-carried time | 90 days
  the number of days before drain removal
Total cost of treatment | 6 month
  The cost of intervention and management of postoperative complications
Return to normal activity | 3 months
  the number of days required for the patient to return to normal activity
Re-intervention | 6 months
  The number of procedures per patient
Hospital stays | 6 months
  the number of admission in the hospital
Patient quality of life | 6 months
  the patient satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed A. Omar, Ass. prof., Principal Investigator — Faculty of medicine, South Valley University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Omar MA, Kamal A, Redwan AA, Alansary MN, Ahmed EA. Post-cholecystectomy major bile duct injury: ideal time to repair based on a multicentre randomized controlled trial with promising results. Int J Surg. 2023 May 1;109(5):1208-1221. doi: 10.1097/JS9.0000000000000403. PMID 37072143